CLINICAL TRIAL: NCT07135297
Title: Novel Thin Bronchoscope Versus Ultrathin Bronchoscope for the Diagnosis of Peripheral Pulmonary Nodules: A Multicenter, Randomised Trial
Brief Title: Novel Thin Bronchoscope Versus Ultrathin Bronchoscope for the Diagnosis of Peripheral Pulmonary Nodules
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Chief Physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IS25002
Record Dates: First submitted 2025-07-22; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer (Diagnosis)
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UTB-VBN-EBUS (Experimental): An ultrathin bronchoscope with an outer diameter of 3.0mm and a working channel of 1.7mm will be used in combination with VBN and EBUS. An outer diameter 1.5mm biopsy forceps and a 1.4mm cytology brush will be used for sample collection.
  Interventions: Device: Ultrathin bronchoscope (UTB)
- TB1-VBN-EBUS-GS (Experimental): A thin bronchoscope with an outer diameter of 3.3mm and a working channel of 2.0mm will be used in combination with VBN and EBUS. A guide sheath with an outer diameter of 1.95mm, a 1.5mm biopsy forceps, and a 1.4mm cytology brush will be used for sample collection.
  Interventions: Device: Thin bronchoscope (TB1)
- TB2-VBN-EBUS-GS (Experimental): A thin bronchoscope with an outer diameter of 4.2mm and a working channel of 2.8mm will be used in combination with VBN and EBUS. A guide sheath with an outer diameter of 2.55mm, a 1.9mm biopsy forceps, and a 1.8mm cytology brush will be used for sample collection.
  Interventions: Device: Thin bronchoscope (TB2)

INTERVENTIONS:
Device: Ultrathin bronchoscope (UTB) — A UTB will be used to perform white light bronchoscopy, then the rEBUS probe was inserted into the working channel and advanced to the PPL to obtain a rEBUS view per the navigation path created by VBN workstation. The probe will be withdrawn from the working channel when an optimal rEBUS view obtained. A 1.5-mm biopsy forceps and 1.4-mm cytology brush will be used to collect samples through the working channel.
  Arms: UTB-VBN-EBUS
Device: Thin bronchoscope (TB1) — A thin bronchoscope will be used to perform white light bronchoscopy. A biopsy kit, including a 1.95-mm outer diameter guide sheath, 1.5-mm biopsy forceps, and 1.4-mm cytology brush, will be used to obtain samples with the guidance of VBN.
  Arms: TB1-VBN-EBUS-GS
Device: Thin bronchoscope (TB2) — A thin bronchoscope will be used to perform white light bronchoscopy. A biopsy kit, including a 2.55-mm outer diameter guide sheath, 1.9-mm biopsy forceps, and 1.8-mm cytology brush, will be used to obtain samples with the guidance of VBN.
  Arms: TB2-VBN-EBUS-GS

SUMMARY:
This is a prospective, randomised, non-inferior, multicenter study in consecutive patients with solid or sub-solid PPLs 8 to 30 mm in diameter.The subjects will be randomly assigned in a 1:1:1 ratio to the 3.0mm outer diameter/1.7mm forceps channel ultrathin bronchoscope group (UTB-VBN-EBUS group), the 3.3mm outer diameter/2.0mm forceps channel novel thin bronchoscope combined with guide sheath group (TB1-VBN-EBUS-GS group), and the 4.2mm outer diameter/2.8mm forceps channel novel thin bronchoscope combined with guide sheath group (TB2-VBN-EBUS-GS group). All procedures will be performed using UTB or TB with the guidance of virtual bronchoscopic navigation (VBN) combined with radial endobronchial ultrasound (rEBUS), but without fluoroscopy. A small forceps will be used in UTB-VBN-EBUS group and TB1-VBN-EBUS-GS group, while a standard forceps will be used in TB2-VBN-EBUS-GS group. Primary endpoint is the diagnostic yield.

DETAILED DESCRIPTION:
This is a prospective, randomised, non-inferior, multicenter study. The inclusion criteria are patients whose chest imaging shows suspiciously malignant peripheral lung nodules (the nodules are surrounded by lung tissue and are located below the segmental bronchus), and the diameter of the lesion is between 8mm and 30mm. The subjects will be randomly assigned in a 1:1:1 ratio to the 3.0mm outer diameter/1.7mm forceps channel ultrathin bronchoscope group (UTB-VBN-EBUS group), the 3.3mm outer diameter/2.0mm forceps channel novel thin bronchoscope combined with guide sheath group (TB1-VBN-EBUS-GS group), and the 4.2mm outer diameter/2.8mm forceps channel novel thin bronchoscope combined with guide sheath group (TB2-VBN-EBUS-GS group). All procedures were performed using UTB or TB with the guidance of virtual bronchoscopic navigation (VBN) combined with radial endobronchial ultrasound (rEBUS), but without fluoroscopy. A small forceps was used in UTB-VBN-EBUS group and TB1-VBN-EBUS-GS group, while a standard forceps was used in TB2-VBN-EBUS-GS group. Primary endpoint is the diagnostic yield. The secondary endpoints include total examination time, the time from bronchoscope insertion of the glottis to the time of removing from the glottis; duration time of finding lesions, the time from insertion of ultrasound probe to withdrawal of ultrasound probe when a rEBUS view was seen; the proportion of lesions visible by rEBUS; factors affecting the diagnostic yield, difference in the bronchus level reached with the bronchoscope; difference in diagnostic yield; and complication rate. Complication rate includes adverse events related to the procedure during or within 1 month after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Chest imaging shows the presence of peripheral pulmonary lesions (defined as those lesions that are surrounded by pulmonary parenchyma and located below the segmental bronchus) that need to be confirmed by pathology. The length diameter of the lesion is no less than 8 mm and no more than 30mm.
* Patients without contraindications of bronchoscopy.
* Patients have good medical adherence and signed informed consent.

Exclusion Criteria:

* Peripheral pulmonary lesion is pure ground-glass opacity.
* Visible lumen lesions in segment and above segment bronchus during bronchoscopy (evidence of endobronchial lesion, extrinsic compression, submucosal tumor, narrowing, inflammation or bleeding of the bronchus).
* The target lesion has been treated.
* Diffuse pulmonary lesions.
* The investigators believe that patient has other conditions that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | up to 6 months
  Diagnostic yield of ultrathin and thin bronchoscope for peripheral pulmonary nodules

SECONDARY OUTCOMES:
Total examination time | During the procedure
  Total examination time is defined from the time that the bronchoscope is inserted beyond the glottis, until the bronchoscope has been removed from the glottis after examination
Duration of finding lesions | During the procedure
  Duration of finding lesions defined from insertion of ultrasound probe to withdrawal of ultrasound probe
Factors affecting the diagnosis yield | Up to 6 months
  The factors affecting the diagnostic yield includes the nodules nature, size, location, the position of the ultrasound probe relative to the lesions etc.
Difference in the bronchus level reached with the bronchoscope | During the procedure
  Level: Bronchus is level 0, leaf bronchus is level 1, segment bronchus is level 2, sub-segment bronchus is level 3, and so on, such as: LB3a is level 3
Difference in diagnostic yield between the two novel thin bronchoscopes groups | Up to 6 months
  Difference in diagnostic yield between the two novel thin bronchoscopes with guide sheath combined small biopsy forceps and conventional biopsy forceps.
Complication rate | 1 month
  The complications refer to the total of serious adverse events related to the procedure during or within 1 month after the operation.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Shanghai Chest Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asano F, Shinagawa N, Ishida T, Shindoh J, Anzai M, Tsuzuku A, Oizumi S, Morita S. Virtual bronchoscopic navigation combined with ultrathin bronchoscopy. A randomized clinical trial. Am J Respir Crit Care Med. 2013 Aug 1;188(3):327-33. doi: 10.1164/rccm.201211-2104OC. PMID 23600452
- [Background] Oki M, Saka H, Ando M, Asano F, Kurimoto N, Morita K, Kitagawa C, Kogure Y, Miyazawa T. Ultrathin Bronchoscopy with Multimodal Devices for Peripheral Pulmonary Lesions. A Randomized Trial. Am J Respir Crit Care Med. 2015 Aug 15;192(4):468-76. doi: 10.1164/rccm.201502-0205OC. PMID 26039792
- [Background] Oki M, Saka H, Asano F, Kitagawa C, Kogure Y, Tsuzuku A, Ando M. Use of an Ultrathin vs Thin Bronchoscope for Peripheral Pulmonary Lesions: A Randomized Trial. Chest. 2019 Nov;156(5):954-964. doi: 10.1016/j.chest.2019.06.038. Epub 2019 Jul 26. PMID 31356810
- [Background] Asano F, Ishida T, Shinagawa N, Sukoh N, Anzai M, Kanazawa K, Tsuzuku A, Morita S. Virtual bronchoscopic navigation without X-ray fluoroscopy to diagnose peripheral pulmonary lesions: a randomized trial. BMC Pulm Med. 2017 Dec 11;17(1):184. doi: 10.1186/s12890-017-0531-2. PMID 29228929
- [Background] Yoshikawa M, Sukoh N, Yamazaki K, Kanazawa K, Fukumoto S, Harada M, Kikuchi E, Munakata M, Nishimura M, Isobe H. Diagnostic value of endobronchial ultrasonography with a guide sheath for peripheral pulmonary lesions without X-ray fluoroscopy. Chest. 2007 Jun;131(6):1788-93. doi: 10.1378/chest.06-2506. PMID 17565021
- [Background] Steinfort DP, Khor YH, Manser RL, Irving LB. Radial probe endobronchial ultrasound for the diagnosis of peripheral lung cancer: systematic review and meta-analysis. Eur Respir J. 2011 Apr;37(4):902-10. doi: 10.1183/09031936.00075310. Epub 2010 Aug 6. PMID 20693253
- [Background] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779